CLINICAL TRIAL: NCT03453931
Title: Arrhythmias, Heart Rate Variability and Microalbuminuria After Intravenous Corticosteroids: An Observational Study
Brief Title: Arrhythmias, Microalbuminuria and Corticosteroids
Status: Completed | Type: Observational
Sponsor: Elza Abdessater (Other)
Responsible Party: Sponsor-Investigator, Elza Abdessater, Medical Student (Master 4), Université Libre de Bruxelles
Organization: Université Libre de Bruxelles (Other)
Other Study IDs: P2017/556 / B406201734265
Record Dates: First submitted 2018-02-10; First posted 2018-03-05 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Corticosteroids Adverse Reaction
Keywords: Corticosteroids; Arrhythmia; Heart Rate Variability; Albuminuria
MeSH Terms: conditions — Arrhythmias, Cardiac; Albuminuria | interventions — Adrenal Cortex Hormones; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Corticosteroid injection — Intravenous high dose corticosteroids
  Other Names: Solumedrol

SUMMARY:
The goal of this observational design is to study the effects of intravenous corticosteroids on heart rate variability, arrhythmias and microalbuminuria. Some previous studies have shown that intravenous corticosteroids could induce bradycardia but also supra-ventricular tachycardia and atrial fibrillation.

A second goal of this study is to investigate whether exogenous corticosteroids may induce microalbuminuria. A large retrospective study has revealed an association between microalbuminuria and corticosteroid use in the year preceding the measurement.

DETAILED DESCRIPTION:
On intra-hospital patients, it will be explored the prevalence of arrythmias, the heart rate variability and the modification of the microalbuminuria level after intravenous infusion of corticosteroids. The investigator shall not initiate the treatment. Patients will receive high-dose intravenous corticosteroids for the treatment of different diseases. The departments, where the patients are enrolled, are: nephrology, neurology, dermatology and rheumatology and the day hospital. The day before the corticosteroids administration, a holter monitor will be started for at least 24h to detect arrhythmias and heart rate variations. By mean of a Finometer, beat-to-beat blood pressure, cardiac output and baroreflex sensitivity will be measured before, during and after the infusion. Blood and urine samples will be used to explore the effects of corticosteroids on microalbuminuria, electrolytes, CRP and glomerular filtration rate during the 3 days of observation.

To our knowledge, it will be the first prospective trial to explore a link between intravenous corticosteroids administration and heart rate variability, Baroreflex Sensitivity, as well as microalbuminuria.

ELIGIBILITY:
Inclusion Criteria:

* Starting high-dose intravenous corticotherapy

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients who are starting high-dose corticotherapy in Hôpital Erasme (Brussels).
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Arrhythmias | Change between day 1 and day 3
  All types of arrhythmias (especially pauses and atrial fibrillation). Evaluated with a 72-hours Holter ECG monitoring
Microalbuminuria | Change in microalbuminuria (day 1 and day 3)
  Microalbuminuria (mg/dL)
Microalbuminuria - Urinary Creatinine ratio | Change in microalbuminuria - urinary creatinine ratio (day 1 and day 3)
  mg/g creatinine

SECONDARY OUTCOMES:
Baroreflex Sensitivity | Change in Baroreflex Sensitivity (day 1 and day 3)
  Measured with a Finometer (ms/mmHg)
Beat-to-beat blood pressure | Change in beat-to-beat blood pressure (day 1 and day 3)
  Measured with a Finometer (mmHg)
Heart Rate | Change in Heart Rate (day 1 and day 3)
  Measured with a 72 hours Holter ECG monitoring (bpm)
Standard Deviation of normal to normal R-R intervals (SDNN) | Change in SDNN (day 1 and day 3)
  Measured with a 72 hours Holter ECG monitoring (ms)
Root Mean Square of the Successive Differences (RMSSD) | Change in RMSSD (day 1 and day 3)
  Measured with a 72 hours Holter ECG monitoring (ms)
Mean number of times per hour in which the change in consecutive normal sinus R-R intervals exceeds 50 milliseconds (PNN50) | Change in PNN50 (day 1 and day 3)
  Measured with a 72 hours Holter ECG monitoring (%)
Low Frequency component of Heart Rate Variability (LF) | Change in low frequencies (day 1 and day 3)
  Measured with a 72 hours Holter ECG monitoring (ms^2)
High Frequency component of Heart Rate Variability (HF) | Change in high frequencies (day 1 and day 3)
  Measured with a 72 hours Holter ECG monitoring (ms^2)
Low to High Frequency Ratio of Heart Rate Variability (LF/HF) | Change in LF/HF (day 1 and day 3)
  Measured with a 72 hours Holter ECG monitoring

OTHER OUTCOMES:
CRP | before and 1 to 3 days after the drug infusion
  (mg/L)
Glomerular Filtration Rate | Before and 1 to 3 days after the drug infusion
  CKD-EPI (mL/min/1.73m2)
Natremia | Change in Natremia (day 1 and day 3)
  mmol/L
Kaliemia | Change in Kaliemia (day 1 and day 3)
  mmol/L
Chloremia | Change in Chloremia (day 1 and day 3)
  mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Marc Leeman, PhD, Study Director — Université Libre de Bruxelles
Locations (1):
- Erasme hospital, Brussels, Belgium